CLINICAL TRIAL: NCT03526952
Title: An Internet Delivered Intervention for Re-Adjustment to Sexual Intimacy With an Ostomy After Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); York University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 352-2016
Record Dates: First submitted 2018-04-10; First posted 2018-05-16 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer; Sexual Dysfunction
MeSH Terms: conditions — Colorectal Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Couples in this group will receive the Internet-Delivered Intervention for Sexual Re-Adjustment
  Interventions: Other: Internet-Delivered Intervention for Sexual Re-Adjustment
- Educational Comparison Group (Active Comparator): Couples in this group will receive only written educational material about sexuality and intimacy with an ostomy.
  Interventions: Other: Written Educational Material

INTERVENTIONS:
Other: Internet-Delivered Intervention for Sexual Re-Adjustment — Couples will meet with a therapist via video-conferencing for two 1.5-hr sessions. The therapist will facilitate couples' communication about their sexual and intimate relationship while providing psychoeducation about couple coping and sexuality after cancer and with an ostomy. Discussion will focus on current concerns, motivations for sex, relational strengths, and intimacy and sensual pleasure. Couples will also be encouraged to practice a sensate focusing exercise between sessions.
  Arms: Intervention Group
Other: Written Educational Material — Couples will receive written educational material for patients coping with changes in intimacy and sexuality when living with a permanent ostomy. This educational material is published by the United Ostomy Associations of America, Inc. and is available for free download from their website. Couples will have two weeks to read this material.
  Arms: Educational Comparison Group

SUMMARY:
This study investigates the feasibility and efficacy of an Internet-delivered intervention for the sexual and intimate re-adjustment of couples in which one partner is living with a temporary or permanent ostomy (e.g., colostomy, ileostomy, urostomy) following treatment for colorectal and/or bladder cancer. The two session intervention will be delivered via online videoconferencing and will focus on facilitating couples' communication around their sexual and intimate relationship. Exercises from sex therapy will be used to scaffold conversations about motivations for having sex, intimacy and sensual pleasure, and relational strengths for coping. The intervention aims to enhance couples' ability to cope with the changes in their sexual and intimate relationship. A group of couples receiving written educational material only will be used as a comparison group to measure change in sexual and intimate adjustment over time.

ELIGIBILITY:
Inclusion criteria:

Patients meeting all of the following criteria will be eligible for the study:

* Patients who have had a diagnosis of colorectal and/or bladder cancer within their lifetime
* Patients who are at least 1-month post active treatment for colorectal and/or bladder cancer
* Patients who have an ostomy due to colorectal and/or bladder cancer (e.g., colostomy, ileostomy, urostomy; permanent or temporary)
* Patients who are in a committed intimate relationship
* Patients who report changes in their sexual/intimate relationship associated with colorectal and/or bladder cancer and/or living with an ostomy
* Patients who have access to the Internet in a private space
* Patients who reside in Ontario
* Patients who are 18 years of age or older

OR

Partners of patients who meet the above criteria and who are 18 years of age or older

Exclusion criteria:

Patients/couples will be excluded from study participation if:

* Patient is undergoing active treatment for cancer
* Patient or partner report high levels of relational distress and would be better suited to couples therapy
* Couple is attending or plans to attend couples or sex therapy concurrently with participation in study
* Patient or partner is currently experiencing mental health concerns that would interfere with study participation (e.g., suicidal ideation, psychotic disorders, substance abuse, spousal abuse)
* Patient or partner lack English proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in sexual functioning from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Sexual Functioning Questionnaire (SFQ): A measure sexual functioning developed specifically for cancer patients and their partners. This measure includes 22 scored items and nine subscales related to different areas of concern (i.e., Interest, Desire, Arousal, Satisfaction, Activity, Orgasm, Masturbation, Relationship, and Problems). For these subscales, higher scores represent better functioning. The optional 5-item Health Impact Scale assess the impact of cancer on the patient's sexual functioning and can be adapted for the partner. For the Health Impact subscale, higher scores represent greater impact.
Change in communication about sex from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Dyadic Sexual Communication Scale (DSC): The DSC scale is a 13-item scale that measures how respondents perceive the discussion of sexual matters with their partners. Items are rated on a 6-point Likert type scale (1 = Disagree Strongly, 6 = Agree Strongly).
Change in perceived self efficacy in coping with sexual and intimate changes from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Sexual Self-Efficacy: A 3-item questionnaire for assessing individual's perceived self-efficacy in coping with sexual and intimate change in the context of cancer. Respondents rate their level of confidence in coping with these changes on a scale of 0-100 (0 = cannot do at all, 100 = highly certain can do).
Change in relational identity or closeness from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  "We-ness" Questionnaire: A measure of the degree partner's perceive themselves more as being a unit ("we/us") than two separate identities ("I/me" or "you/him/her"), which encompassed an intertwined structure of affective, cognitive, and behavioural facets. The questionnaire includes 16-items about facets of couples' mutual identity and respondents use a 5-point Likert scale to rate the degree to which these facets contribute to their sense of mutual identity in their current relationship. Higher scores represent a greater sense of shared identity.
Change in mutual identity from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Inclusion of Other In Self Scale (IOSS): The IOSS is a one-item, visual measure of the degree to which one views one's partner as being part of one's self-concept. Respondents choose one of seven Venn-diagram type images that represent varying degrees of mutual identity. Higher scores represent greater degrees of self-other overlap in identity.

SECONDARY OUTCOMES:
Change in relational adjustment from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Revised Dyadic Adjustment Scale: A 14-item self-report questionnaire measuring respondents' relational adjustment in terms of consensus, satisfaction, and cohesion. Items are scaled on a 6-point Likert scale.
Change in psychological adjustment (depression) from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Centre for Epidemiological Studies Depression Scale- Revised (CESD-R): A brief 20-item self-report measure of depressive symptoms experienced over the past week. Respondents indicate how often they have experienced the symptoms over the past week using a 5-point Likert scale. Higher scores indicate higher risk for clinical depression.
Change in psychological adjustment (anxiety) from four different time points | This questionnaire will be completed by participants at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Generalized Anxiety Disorder-7 (GAD-7): A brief, 7-item, self-report measure of generalized anxiety. Respondents indicate how often they have experienced symptoms of generalized anxiety over the past two weeks, using a 4-point Likert scale. Higher scores indicate greater levels of difficulty.
Patients' change in adjustment to colorectal cancer from four different time points | This questionnaire will be completed by patients diagnosed with colorectal cancer at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Functional Assessment for Cancer Treatment - Colorectal Cancer (FACT-C): The "Colorectal Cancer" subscale of the FACT-C will be completed by patients only as a measure of their adjustment to the colorectal cancer and ostomy. The subscale includes 9-items about physical and psychological symptoms related to colorectal cancer and respondents are to indicate the degree to which they experienced these symptoms in the past week using a 5-point Likert scale (0 = not at all, 5 = very much).
Patients' change in adjustment to bladder cancer from four different time points | This questionnaire will be completed by patients diagnosed with bladder cancer at T0 (baseline), T1 (within 1-week after intervention), T2 (1-month after intervention), and T3 (3-months after intervention)
  Functional Assessment for Cancer Treatment - Bladder Cancer (FACT-Bl): The "Bladder Cancer" subscale of the FACT-Bl will be completed by patients only as a measure of their adjustment to the colorectal cancer and ostomy. The subscale includes 9-items about physical and psychological symptoms related to bladder cancer and respondents are to indicate the degree to which they experienced these symptoms in the past week using a 5-point Likert scale (0 = not at all, 5 = very much).

OTHER OUTCOMES:
Expectancy for Change | This questionnaire will be completed once at T0 (baseline)
  Credibility/expectancy questionnaire: A brief 6-item measure of treatment expectancy and rationale credibility.
Therapeutic Alliance | This questionnaire will be completed once at T1 (within 1-week after intervention)
  Working Alliance Inventory Short Form-Revised (WAI-SR): The WAI-SR will be used to measure each participant's working alliance with the therapist facilitating the two session intervention. The WAI-SR is a 12-item self-report measure of working alliance from the client's perspective that uses a 5-point Likert scale, where higher score represent better working alliance between client and therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fergus, PhD, C.Psych, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The study will be shared via publication(s) in an academic journal and/or conference presentation(s)